CLINICAL TRIAL: NCT07280364
Title: Metabolomics in the Diagnosis and Treatment of Asthma in Children
Status: Recruiting | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 03-24
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Asthma
Keywords: bronchial asthma; children; metabolomics; metabolites
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Standart medical treatment — No intervention, patients will recieve standard medical treatment

SUMMARY:
The goal of this observational study is to learn about the metabolomic profile of blood and urine in children 12-17 years with asthma. The main question it aims to answer is:

• Are there metabolites in the blood and urine that are specific for asthma exacerbation? Participants already receive standard therapy as part of their regular medical care for asthma.

DETAILED DESCRIPTION:
The study plans to enroll 100 children with a confirmed diagnosis of bronchial asthma of varying severity. Patients will be divided into groups based on disease severity (mild and severe/moderate) and stage (exacerbation/non-exacerbation). A separate group of patients receiving targeted therapy will also be included. All patients will be hospitalized in the pulmonology department. Blood and urine samples will be collected for metabolomic analysis upon admission. Patients not experiencing an exacerbation will not be re-evaluated. For patients experiencing an asthma exacerbation, blood and urine samples will be collected again after 10 days. Throughout the study, patients will receive the usual therapy prescribed by their treating physician. Treatment for exacerbations includes inhaled budesonide and ipratropium bromide/fenoterol via a nebulizer; systemic steroids may be used if indicated. All patients will undergo spirometry upon admission to the department. Patients in the acute stage will undergo spirometry at least twice, including on the 10th day, plus or minus 2 days. All patients complete the Asthma Control Test questionnaire upon admission.

ELIGIBILITY:
Inclusion Criteria:

* Age from 12 to 17 years old
* Confirmed diagnosis of asthma
* Informed voluntary consent to participate in the study

Exclusion Criteria:

* age under 12 years
* no established diagnosis of asthma
* concomitant severe somatic, metabolic, and endocrine diseases
* patient's withdrawal of informed consent

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will include children hospitalized in the pulmonology department of the Sechenov Center for Maternity and Childhood Care at Sechenov University.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
inflammation biomarkers | baseline and 10 days
  Identification of metabolomic changes (inflammation biomarkers) in the blood (aminoacids) and urine (organic acids) of patients with mild, moderate, and severe bronchial asthma associated with asthma exacerbation.

SECONDARY OUTCOMES:
metabolomic changes | baseline and 10 days
  Changes in the metabolomic profile of blood and urine depending on the severity of asthma and the therapy being administered: compare the urine metabolomic profile for organic acids and aminoacids in blood in children with mild and modereate/severe asthma. Assess the dynamics of blood and urine metabolomic profiles in children with severe asthma before and after therapy with biologic agents.Identify the relationship between the blood and urine metabolomic profile in children with asthma and respiratory function parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia A. Geppe, MD, Doctor of M.Sc., Professor, Principal Investigator — I.M. Sechenov First Moscow State Medical University
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No